CLINICAL TRIAL: NCT02345759
Title: Psychological Aspects Related to Compliance of Patients on Restricted-protein Regimens in Chronic Kidney Disease
Brief Title: Psychological Aspects and Patients Compliance to Restricted-protein Regimens in Chronic Kidney Disease
Acronym: KetoPsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Sponsor
Other Study IDs: AWG 5/2014
Record Dates: First submitted 2014-08-23; First posted 2015-01-26 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Psychological Characteristics Involved in Dietary Compliance
Keywords: CKD patients; protein-restricted diets; compliance; psychological aspects
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Keto-diet group: Vegetarian very low protein regimen (0.3 g proteins/kg ideal body weight per day) supplemented with ketoanalogues of essential amino acids (Ketosteril®, Fresenius Kabi, Bad Homburg, Germany), 1 capsule for every 5 kg of ideal dry body weight per day.
- Conventional LPD group: 0.6 g/kg per day, including high biological value proteins

SUMMARY:
Dietary management of CKD patients proved important to postpone dialysis. Long-term compliance to protein-restricted diets was discussed. Psychological aspects involved in certain dietary behaviour have never been studied.

DETAILED DESCRIPTION:
The interest in dietary management resurged, since the high prevalence of revealed a major impact not only on morbidity, mortality, social activities and patients' quality of life, but also on health budget.

Although protein-restricted diets are used for more than a century in patients with advanced Chronic Kidney Disease (CKD), their efficacy and safety is still debatable. Enough evidence has being accumulated on their role in postponing dialysis initiation in compliant patients. Consequently, the long-term compliance to the diet is discussed. Psychological aspects of compliant patients are certainly involved. Identification of certain psychological predictors of dietary compliance could help to select the patients who are more likely to be compliant and therefore to benefit from such an intervention. Moreover, short-term or long-term psychological intervention addressing these factors could increase patient long-term compliance.

Accordingly, we are aiming to evaluate psychological characteristics of Chronic Kidney Disease patients in relation with their compliance to protein-restricted regimens.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* stage 4+ CKD
* good nutritional status (Subjective Global Assessment score A/B and serum albumin ≥3.5 g/dL)
* declared potentially good compliance with a low protein diet and agreed to follow the monitoring schedule are considered for the program

Exclusion Criteria:

* poorly controlled arterial blood pressure (≥145/85 mm Hg)
* uncontrolled diabetes mellitus
* other relevant comorbidities (heart failure, active hepatic disease, digestive diseases with malabsorption, inflammation/anti-inflammatory therapy)
* uremic complications (pericarditis, polyneuropathy)
* feeding inability (anorexia, nausea)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients, with stage 4-5ND CKD (estimated glomerular filtration by MDRD formula of less than 30 mL/min per year) included in the dietary intervention program of "Dr Carol Davila" Teaching Hospital of Nephrology coming for the scheduled visits between January the 1st and June the 30th, 2014 will be considered eligible.
  Those who will sign the informed consent will be included in the study; the specially-designed questionnaire will be administered. Simultaneously, their routine assesment, including the dietary compliance, manifestations of CKD and the nutritional status will be performed, as recommended by the Romanian Best Practice Guidelines for CKD [28].
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Compliance to the protein-restricted diet | 12 months
  The compliance to the diet is appreciated to be good if both the achieved protein intake and the achieved energy is in the range of ±10% of the recommended values.

SECONDARY OUTCOMES:
Parameters related to renal function (The decline in glomerular filtration rate (GFR) GFR decline | 12 months
  The decline in glomerular filtration rate (GFR)
Psychological parameter - self-efficacy score | 12 months
  Self-efficacy score derives from the self-efficacy scale.
Nitrogen balance (Serum urea level) | 12 months
  Serum urea level
Metabolic acidosis (Serum bicarbonate level) | 12 months
  Serum bicarbonate level
Calcium-phosphorus metabolism abnormalities (Serum calcium) | 12 months
  Serum calcium
Calcium-phosphorus metabolism abnormalities (Serum phosphates level) | 12 months
  Serum phosphates level
Psychological parameter - illness perception (Sub-scores derived from illness perception questionnaire) | 12 months
  Sub-scores derived from illness perception questionnaire: the higher this score, the worse is patient's perception on the disease.
Mental status - vitality index | 12 months
  Vitality score derived from mental component of SF-36
Psychological parameter -mental score | 12 months
  The mental score looks at depression. Psychological difficulties interfere with the initiation of compliance behaviours.

OTHER OUTCOMES:
Safety parameters (Subjective Global Assessment, anthropometric markers, biochemical parameters, and serum total cholesterol) | 12 months
  Parameters of nutritional status are predefined as safety parameters. Subjective Global Assessment anthropometric markers, and biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Professor of Nephrology, Study Chair — Spitalul Clinic de Nefrologie "Dr Carol Davila"; Liliana Garneata, MD, PhD, Study Director — Spitalul Clinic de Nefrologie "Dr Carol Davila"; Cristina Drugau, MD, Principal Investigator — Spitalul Clinic de Nefrologie "Dr Carol Davila"; Evy Dehelean, Psychologist, Principal Investigator — International Health Care Systems Romania
Locations (1):
- Spitalul Clinic de Nefrologie "Dr Carol Davila", Bucharest, Romania